CLINICAL TRIAL: NCT05923788
Title: T1 Mapping in Diagnosis and Follow up of Fabry Disease
Brief Title: T1 Mapping in Fabry Disease
Acronym: MAP-FAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0934; 2023-A00475-40 (Other: ID-RCB)
Record Dates: First submitted 2023-05-24; First posted 2023-06-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; T1 mapping; functional MRI; Fabry nephropathy
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fabry disease (Other)
  Interventions: Diagnostic Test: T1 mapping measurement
- Patients undergoing renal functional exploration (Other): Patients undergoing renal functional exploration for a reason other than Fabry disease, amyloidosis, hemochromatosis
  Interventions: Diagnostic Test: T1 mapping measurement

INTERVENTIONS:
Diagnostic Test: T1 mapping measurement — T1 mapping values to test the ability of the MRI sequence to detect Gb3 in kidney

SUMMARY:
Fabry disease (OMIM-301500, FD) is a lysosomal storage disease with X-linked inheritance secondary to mutations in the α-galactosidase A gene (GLA), which cause absence or decreased activity of the lysosomal hydrolase a-galactosidase A (a-gal A). The accumulation of globotriaosylceramide (Gb3) leads to multiple organs dysfunction, especially in three key organs: kidney, heart and cerebrovascular system. Progressive nephropathy is one of the main features of Fabry disease and is marked by an insidious development. The investigators are facing different current challenges about treatment initiation in non-classic phenotype patients, optimal dose after treatment initiation, and treatments monitoring in Fabry nephropathy. That is even more important that the enzyme replacement therapy is expensive and a lifelong commitment.

Functional magnetic resonance imaging (MRI) is now able to provide T1 mapping sequence. In Fabry disease, T1 mapping is currently used to assess the degree of myocardial involvement. The MRI for assessement of Fabry Cardiomyopathy is now recommended by the 2022 national diagnostic and care protocol (PNDS) in France. However there is no data about T1 mapping values in kidney in Fabry's disease The main Objective is to describe renal performance through multi-parametric MRI in Fabry nephropathy and the primary outcome will be the quantification of renal T1 in Fabry patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed Fabry disease Or Control patients: Patients undergoing renal functional exploration for a reason other than Fabry disease, amyloidosis, hemochromatosis
* Adult patient
* Patient informed of the study and agree to participate
* Patient affiliated to a social security or beneficiaries of a similar scheme

Exclusion Criteria:

* Weight > 130 kg
* kidney transplant,
* polycystic kidney disease,
* Pregnant, parturient or breastfeeding
* Contraindications to MRI
* Subject participating in another research including an exclusion period still in progress at inclusion
* Persons deprived of their liberty by a judicial or administrative decision,
* Adults subject to a legal protection measure (safeguard measure, guardianship, curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
T1 value measured | Day 1
  Difference in the measurement of T1 mapping by MRI in Fabry disease patients compared with controls.
  T1 mapping is a MRI sequence to estimate renal fibrosis

SECONDARY OUTCOMES:
Apparent diffusion coefficient (ADC) coefficient values | Day 1
  ADC coefficient values to measure the degree of fibrosis in Fabry nephropathy in Fabry disease patients compared with controls.
R2* coefficient values | Day 1
  R2* values to measure the degree of renal alteration in Fabry nephropathy in Fabry disease patients compared with controls.
T2 value measured | Day 1
  Comparison of T2 values measured by T2 mapping MRI between patients with Fabry disease and controls.
  T2 mapping is a MRI sequence to estimate renal alteration
T1 mapping measurement Fabry disease | Day 1
  Comparison of T1 mapping values within 3 different subgroups of patients with Fabry disease (treated men, treated or untreated women)
In Fabry disease patients, evaluation of the association between the T1 values measured and concentration of plasma globotriaosylsphingosine (LysoGb3) | Day 1
In Fabry disease patients, evaluation of the association between glomerular filtration rate and ADC value measured | Day 1
  ADC value measured by diffusion-weighted MRI
In Fabry disease patients, evaluation of the association between glomerular filtration rate and R2* value measured | Day 1
  R2* value measured by blood oxygen level-dependent (BOLD) MRI
In Fabry disease patients, evaluation of the association between glomerular filtration rate and T2 value measured | Day 1
  T2 value measured by T2 mapping MRI
In Fabry disease patients, evaluation of the association between proteinuria and ADC value measured | Day 1
  ADC value measured by diffusion-weighted MRI
In Fabry disease patients, evaluation of the association between proteinuria and R2* value measured | Day 1
  R2* value measured by BOLD MRI
In Fabry disease patients, evaluation of the association between proteinuria and T2 value measured | Day 1
  T2 value measured by T2 mapping MRI

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Edouard Herriot, Lyon, France
  - Hopital Femme Mère Enfant, Bron

IPD SHARING:
Plan to Share IPD: No